CLINICAL TRIAL: NCT00154414
Title: Effect of Liraglutide on Glycaemic Control in Japanese Subjects With Type 2 Diabetes.
Brief Title: Effect of Liraglutide on Blood Glucose Control in Japanese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1334; JapicCTI-050131 (Registry Identifier: Japic)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liraglutide

SUMMARY:
This trial is conducted in Japan. The aim of this research trial is to evaluate the effect of treatment with liraglutide or placebo on blood glucose control after 14 weeks in Japanese subjects with type 2 diabetes. Liraglutide or placebo is administered by injection once daily in the evening. The trial is a multi-national trial with treatment concealed to participating subjects, investigators and the sponsor. Treatment allocation is random with equal chance of being assigned to each group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes and treated with diet therapy with or without single oral drug therapy
* 7.0 % =< HbA1c < 10.0 %
* Body Mass Index (BMI) < 30.0 kg/m^2

Exclusion Criteria:

* Subjects treated with thiazolidinediones or insulin
* Subjects with any serious medical conditions

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 14 weeks treatment

SECONDARY OUTCOMES:
Glycaemic control parameters (fasting plasma glucose, post prandial plasma glucose) after 14-week treatment
Body weight after 14 weeks.
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Seino Y, Rasmussen MF, Zdravkovic M, Kaku K. Dose-dependent improvement in glycemia with once-daily liraglutide without hypoglycemia or weight gain: A double-blind, randomized, controlled trial in Japanese patients with type 2 diabetes. Diabetes Res Clin Pract. 2008 Aug;81(2):161-8. doi: 10.1016/j.diabres.2008.03.018. Epub 2008 May 20. PMID 18495285
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com